CLINICAL TRIAL: NCT03024788
Title: Determination of Cut-off Value of Advanced Glycation End-product and Glycosylated Haemoglobin in Type 2 Diabetes Diagnosis in China
Brief Title: Determination of the Optimum Cut-off Value of Type 2 Diabetes Diagnosis Among Chinese Population(SENSIBLE STUDY II)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Zilin Sun, director physician, Zhongda Hospital
Other Study IDs: 2016YFC1305700d
Record Dates: First submitted 2017-01-11; First posted 2017-01-19 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Type II Diabetes
Keywords: Glycosylated haemoglobin; advanced glycation end products
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Syringes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: syringe, fundus camera etc — Physical examination, fundus examination, blood and urine samples collection

SUMMARY:
Study of the correlation between AGEsP and HbA1c and diabetic retinopathy prevalence: determination of cut-off value of AGEsP and HbA1c in type 2 diabetes diagnosis in China

DETAILED DESCRIPTION:
To find the cut-off point of AGEsP and HbA1c for diagnosis of diabetes by drawing the logistic regression model between prevalence of retinopathy and AGEsP level and HbA1c level,and find the point where the prevalence of retinopathy changes most rapidly.

ELIGIBILITY:
Inclusion Criteria:

* 20~70 years old;
* Volunteer to participate in this study and signed informed consent.

Exclusion Criteria:

-

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese natural population
Sampling Method: Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2017-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-12

PRIMARY OUTCOMES:
prevalence of retinopathy | 3 years
  the prevalence of retinopathy in different AGEsP and HbA1c levels

SECONDARY OUTCOMES:
incidence of retinopathy | 3 years
  incidence of retinopathy in different AGEsP and HbA1c levels

IPD SHARING:
Plan to Share IPD: Undecided